CLINICAL TRIAL: NCT06837090
Title: Retrospective Analysis of the Experience With Larotrectinib in Patients With Solid Neoplasms With NTRK Fusion in Spain (SPAINTRK)
Acronym: SPAINTRK
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: MFAR (Other); Grupo Español de Tumores Neuroendocrinos y Endocrinos (GETNE) (Unknown)
Responsible Party: Sponsor
Other Study IDs: GETNE S2411; GETNE S2411/ SPAINTRK (Other: GETNE S2411/ SPAINTRK)
Record Dates: First submitted 2025-02-04; First posted 2025-02-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-03

CONDITIONS: Solid Neoplasms With NTRK Fusions
Keywords: neoplasm; NTRK; Larotrectinib
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thyroid cancer patients with solid neoplasms with NTRK fusions.: Thyroid cancer patients with solid neoplasms with NTRK fusions. The study will use secondary data retrieved from each patient's medical records. The clinical history includes all the clinical variables defined to perform the analysis and it is not necessary to access additional sources.
  The assignment of a patient to a specific therapeutic strategy has already been decided in advance by the usual clinical practice of medicine; the decision to prescribe a specific treatment was clearly dissociated from the decision to include a patient in the study. No intervention, neither diagnostic nor follow-up, will be applied to patients other than usual clinical practice. Epidemiological methods will be used to analyze the data collected.

SUMMARY:
SPAINTRK aims to be the first trial in Spain to systematically collect data on outcomes of Spanish patients with solid neoplasms treated with Larotrectinib through the compassionate drug use program, during the time elapsed between the indication approval and the drug commercialization. This will contribute to selection of the best treatment for cancer patients with NTRK fusions, such as Trk inhibitors like Larotrectinib. Since the FDA and the EMA approved the use of Trk inhibitors, like Larotrectinib, there is a new and effective option of treatment for patients with NTRK fusions in solid neoplasms. This observational retrospective study will allow to analyze data of patients treated with Larotrectinib across the country and increase the knowledge on response to rare and different cancers Main objective is describe the effectiveness of Larotrectinib treatment in tumors with NTRK fusion in Spanish patients as a clinical series.

This is an observational retrospective study including thyroid cancer patients with solid neoplasms with NTRK fusions.

The study will use secondary data retrieved from medical records from each patient. The medical records include all the clinical variables defined in order to perform the analysis and it is not necessary to access additional sources.In total, 19 patients diagnosed with solid neoplasms that have been confirmed to bear NTRK fusions in their tumors will be included in the study. It is known that these patients have received the treatment with Larotrectinib in 14 centers in Spain, prior to treatment reimbursement in Spain.

DETAILED DESCRIPTION:
1. Study title Retrospective analysis of the experience with Larotrectinib in patients with solid neoplasms with NTRK fusion in Spain (SPAINTRK)
2. .RATIONALE AND OBJECTIVES SPAINTRK aims to be the first trial in Spain to systematically collect data on outcomes of Spanish patients with solid neoplasms treated with Larotrectinib through the compassionate drug use program, during the time elapsed between the indication approval and the drug commercialization. This will contribute to selection of the best treatment for cancer patients with NTRK fusions, such as Trk inhibitors like Larotrectinib. Since the Food and Drug Administration (FDA) and the European Medicines Agency (EMA) approved the use of Trk inhibitors, like Larotrectinib, there is a new and effective option of treatment for patients with NTRK fusions in solid neoplasms. This observational retrospective study will allow to analyze data of patients treated with Larotrectinib across the country and increase the knowledge on response to rare and different cancers 2.1 Main Objective Description of the effectiveness of Larotrectinib treatment in tumors with NTRK fusion in Spanish patients as a clinical series.

   2.2. Secondary Objectives
   * Describe treatment duration, including dose reductions and interruptions occurred along the treatment with Larotrebtinib, as well as to study the reasons behind those decisions.
   * Study the effectiveness of Larotrebtinib and previous lines of therapy. Identified the line of treatment at which molecular testing for NTRK was performed.
   * Exploration of clinical and/or histological variables related to the effectiveness and tolerability of Larotrectinib treatment.
3. RESEARCH METHODS 3.1. Study design This is an observational retrospective study including thyroid cancer patients with solid neoplasms with NTRK fusions.

   The study will use secondary data retrieved from medical records from each patient. The medical records include all the clinical variables defined in order to perform the analysis and it is not necessary to access additional sources.

   The assignment of a patient to a specific therapeutic strategy has been already decided in advance by the usual clinical practice of medicine; the decision to prescribe a specific treatment was clearly dissociated from the decision to include a patient in the study. No intervention will be applied to patients, either diagnostic or follow-up, other than the usual clinical practice. Epidemiological methods will be used to analyze the data collected.

   3.2. Setting and study population In total, 19 patients diagnosed with solid neoplasms that have been confirmed to bear NTRK fusions in their tumors will be included in the study. It is known that these patients have received the treatment with Larotrectinib in 14 centers in Spain, prior to treatment reimbursement in Spain.

   3.3. Inclusion Criteria Infant and adult patients (all ages). Patients with confirmed diagnosis of solid neoplasms. Patients must have detected NTRK fusions by the following diagnostic methods NGS, fluorescence in situ hybridization (FISH) and/or Immunohistochemistry (IHC).

   Patients must be treated with Larotrectinib under the compassionate use program (before the commercialization) in order to be included in the study.

   Data should be available in order to evaluate effectiveness and consequent follow up.

   3.4. Exclusion Criteria Patients with solid neoplasms treated with Larotrectinib in clinical trials or other settings different from clinical practice.

   Patients that initiated treatment with Larotrectinib after the obtention of prize-reimbursement and commercialization.

   3.5. Study Size The sample size calculation is based on the actual number of patients known to be treated in Spain with Larotrectinib. At the moment 19 patients from 14 different healthcare centers have been localized that were treated in the Spanish territory with Larotrectinib. We expect to include and collect data from all of them.

   3.6. Sampling and recruitment method Patients will be consecutively included, in compliance with the previously established inclusion criteria.

   According to the definition of study population and disease established in this scientific report, patients will be selected from cases diagnosed with solid neoplasms bearing NTRK fusions detected by any of these methods, NGS, FISH and/or IHC, and treated with Larotrectinib. The 19 patients treated with Larotrectinib in the Spanish territory are localized and belong to 14 different sites/healthcare centers.

   To prevent two or more reporting physicians from logging the same case, a coordinator, who controls the cases included in his or her center, is appointed in health centers with several reporting physicians, and preventive measures are implemented in the tool controlling duplications in variables (such as birth date, gender, center or diagnosis).

   3.7. Case Definition A 'case' is defined as any patient, diagnosed, treated, or followed in the different health centers where reporting physicians authorized by the sponsor, who meets the inclusion criteria. A key point is that the patient was diagnosed with solid neoplasms that harbors a NTRK fusion and he/she was receiving treatment with Larotrectinib. Data from patient's treatment should have been recorded and be available at the centers.

   3.8. Data Logging Once the patient is compliant with inclusion/exclusion criteria information on the clinical history will be collected to gather the necessary data and to complete the electronic forms of the study designed for this purpose. All data collected during treatment, as well as demographic data, will be provided for the purpose of this study and completed at the electronic Case Report Form (eCRF) to proceed to its analysis.
4. ENDPOINTS AND VARIABLES 4.1. Endpoints 4.1.1. Primary Endpoints Duration of response (DoR): is defined as the time from first confirmed response (complete (CR) or partial (PR) response), according to Objective response rate (ORR) defined below, to the date of the documented progression of the disease (PD) as determined using RECIST V1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.

   Results will be presented as individual cases, not compiled as the patients have different pathologies which may differ in prognosis.

   4.1.2. Secondary Effectiveness Endpoints
   * Objective response rate (ORR): is assessed by the investigator analysis of tumor growth through imaging follow-up (CT scan/MRI), using a method to evaluate it as RECIST V1.1. This will be considered as the number of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the period of treatment with Larotrectinib. Tumor measurements that were assessed locally by the clinician according to RECIST, V1.1, should be recorded and indicate the change in size of tumors as compared with baseline, at the first dose of study treatment.
   * Progression free survival (PFS): Time from first dosing date to the date of confirmed PD according to RECIST 1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
   * Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patients' status at each visit.

   Results will be presented as individual cases, not compiled as the patients have different pathologies which may differ in prognosis.

   4.1.3. Secondary Safety Endpoints

   -Safety: All safety information will be collected retrospectively according to data available in the chart review. A descriptive analysis of adverse events collected in medical charts will be done taking into account:
   1. The frequency of Adverse events (AEs) will be reported per patient by MedDRA System Organ Class (SOC) and Preferred Term (PT);
   2. The maximum CTCAE grade will be reported per patient;
   3. The causal relationship with the study drug will be assessed locally by the investigator

      - Larotrectinib interruptions / Delays: number of interruptions and delays of treatment reported per patient (frequency) and reason for dose interruption / delay.
      * Larotrectinib dose reductions or modifications: Number of reductions or modifications of doses reported per patient (frequency) and reason for dose reduction / modification.
      * Larotrectinib treatment duration: Time elapsed between first dose and permanent discontinuation of the study treatment.

      4.2. Study Variables

      Investigators will provide information of each of the following variables:

      Variables for Demography:

      - Age at enrollment.
      * Sex (male, female).
      * Race (white, black, Asian, other)
      * Height (cm).
      * Weight (kg).
      * Body mass index.
      * Body surface area (BSA) - calculated from the reported height and weight using Mostseller's formula:

      BSA (m2)= (height (cm) x weight (kg) / 3600) 1/2

      - Performance status.will be presented using the Eastern Cooperative Oncology - Group (ECOG) scale.

      Cancer history:
      * Primary cancer diagnosis.
      * Primary tumor type, histology and location
      * Stage of disease at initial diagnosis(I-IV).
      * Time since initial diagnosis.
      * Extent of disease at enrollment (metastatic, locally advanced, sites of disease, presence of at least one measurable lesion). Stage of the disease at inclusion
      * Time since diagnosis of metastatic or locally advanced disease (years).

      Prior anticancer treatments:

      -Prior systemic treatments type, start and end dates.

      -Number of prior systemic regimens or treatment courses.

      -Best overall response to the most recent prior systemic regimen or treatment course (CR, PR, stable disease, progressive disease, unknown or inevaluable or not applicable).

      -Prior radiotherapy.

      -Prior cancer-related surgery.

      NTRK fusions:

      -NTRK fusion gene: NTRK1, NTRK2, NTRK3.

      -NTRK fusion isoform (i.e ETV6-NTRK3).

      -Method of detection: NGS, FISH or IHC and dates of the determinations.
      * Other oncogenic alterations present.

      Treatment with Larotrectinib:

      -Dose of Larotrectinib.

      -Larotrectinib start and end date. Reasons for end of treatment

      -Data records of dose reductions and/or interruptions and their reason.

      -Best response and best response date

      -Progression date.

      -Frequency of AEs reported per patient by MedDRA System Organ Class (SOC) and Preferred Term (PT); the maximum CTCAE grade will be reported per patient. Causal relationship with the study treatment will be reported for all events.

      Survival:
      * Patient status (alive, death, lost to follow-up)
      * Reasons of death (if applicable)
      * Subsequent anticancer treatments (type, start and end dates, best response, progression dates)

ELIGIBILITY:
Inclusion Criteria:

1. Infant and adult patients (all ages).
2. Patients with confirmed diagnosis of solid neoplasms.
3. Patients must have detected NTRK fusions by the following diagnostic methods NGS, fluorescence in situ hybridization (FISH) and/or Immunohistochemistry (IHC).
4. Patients must be treated with Larotrectinib under the compassionate use program (before the commercialization) in order to be included in the study.
5. Data should be available in order to evaluate effectiveness and consequent follow up.

Exclusion Criteria:

1. Patients with solid neoplasms treated with Larotrectinib in clinical trials or other settings different from clinical practice.
2. Patients that initiated treatment with Larotrectinib after the obtention of prize-reimbursement and commercialization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thyroid cancer patients with solid neoplasms with NTRK fusions.
Sampling Method: Probability Sample
Enrollment: 19 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Duration of response (DoR) | Throughout the study period, an average of 1 year
  Duration of response (DoR): is defined as the time from first confirmed response (complete (CR) or partial (PR) response), according to Objective response rate (ORR) defined below, to the date of the documented progression of the disease (PD) as determined using RECIST V1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
  Results will be presented as individual cases, not compiled as the patients have different pathologies which may differ in prognosis

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, an average of 1 year
  Objective response rate (ORR) is assessed by the investigator analysis of tumor growth through imaging follow-up (CT scan/MRI), using a method to evaluate it as RECIST V1.1. This will be considered as the number of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the period of treatment with Larotrectinib. Tumor measurements that were assessed locally by the clinician according to RECIST, V1.1, should be recorded and indicate the change in size of tumors as compared with baseline, at the first dose of study treatment.
Progression free survival (PFS) | Throughout the study period, an average of 1 year
  Progression free survival (PFS): Time from first dosing date to the date of confirmed PD according to RECIST 1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
Overall survival (OS): | Throughout the study period, an average of 1 year
  Overall survival (OS): defined as the time elapsed from the first dose of study treatment until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patients' status at each visit.
  Results will be presented as individual cases, not compiled as the patients have different pathologies which may differ in prognosis.
Safety_ Frequency of AEs | Throughout the study period, an average of 1 year
  Percentage of patients who experienced AEs
Safety _Toxocities | Throughout the study period, an average of 1 year
  Percentage of patients who experienced treatment related adverse events
Larotrectinib interruptions | Throughout the study period, an average of 1 year
  Percentage of patients with larotrectinib interruptions
Larotrectinib dose reductions | Throughout the study period, an average of 1 year
  Percentage of patients with larotrectinib reductions
Larotrectinib treatment duration | Throughout the study period, an average of 1 year
  Larotrectinib treatment duration. Time elapsed between first dose and permanent discontinuation of the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Hernando Cubero, M.D., Ph.D., Study Director — Hospital Vall d'Hebron
Locations (14):
- Spain (14):
  - Hospital Quirón Salud Torrevieja, Torrevieja, Alicante
  - Hospital Universitario Son Espases, Palma, Baleres
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital San Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizkaia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Clínico Santiago de Compostela, Santiago de Compostela, La Coruña
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Universitario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No